CLINICAL TRIAL: NCT00741065
Title: DESWT-Pilot Study on the Safety of Myocardial Regeneration by Direct Epicardial Shock Wave Therapy in Combination With Coronary Artery Bypass Grafting
Acronym: DESWT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cardiac Regeneration Technologies, LLC (Industry)
Responsible Party: Reiner Schultheiss MD, Cardiac Regeneration Technologies LLC
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DESWT,Version:02; May 21,2008
Record Dates: First submitted 2008-08-25; First posted 2008-08-26 (Estimated); Last update posted 2010-02-11 (Estimated); Status verified 2010-02

CONDITIONS: Reduced Left Ventricular Function Defined as LVEF < 50%; Regional Left Ventricular Wall Motion Abnormalities
Keywords: Coronary Artery Bypass Grafting; Myocardial Regeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Direct Epicardial Shock Wave Therapy — performed in adjunct to a standard coronary artery bypass grafting procedure Prior to aortic cross clamping direct epicardial shock wave therapy - applied directly to the myocardium
  Other Names: CardioGold® CG050: CG05000001; CardioGold® CG050: CG05000002; Applikator CA01

SUMMARY:
Study purpose: To examine the safety of myocardial regeneration by direct epicardial shock wave therapy in combination with coronary artery bypass grafting.

DETAILED DESCRIPTION:
Direct epicardial shock wave therapy: DESWT will be performed in adjunct to a standard CABG procedure. Prior to aortic cross clamping, DESWT will be performed using a CardioGold® CG050 (CRT Cardiac Regeneration Technologies, Woodstock, USA / manufactured by MTS-Europe GmbH, Konstanz, Germany) shock wave therapy device and a specially designed handheld applicator under sterile conditions. Depending on the localisation of the myocardial infarct scar, 290-310 impulses will be applied to the anterior, lateral, or posterior wall. Shock waves will be generated at 1 or 2 Hz in a non ECG triggered fashion, should DESWT result in significant ventricular arrhythmias, ECG gating will be initiated. After completion of DESWT, CABG will be continued in a regular fashion.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients above 18 years of age undergoing primary coronary artery bypass grafting.
* Patients have to present with reduced left ventricular function defined as LVEF < 50%.
* Patients have to present with regional left ventricular wall motion abnormalities.
* Patients have to give written informed consent to participate in the study.

Exclusion Criteria:

* Significant concomitant valve disease(except significant valve disease not detected in preoperative cardiac ultrasound that is detected intra-operatively).
* HIV positive patients.
* Hepatitis C positive patients.
* Patients in cardiogenic shock.
* Patients with a contraindication for cardiac MRI.
* Present contraindication for transoesophageal echocardiography (TEE).
* History of significant ventricular arrhythmias, except arrhythmias associated with MI.
* Highly reduced left ventricular function defined as LVEF <30%.
* Present co-morbidity which reduces life expectancy to less than 6 months.
* Presence of ventricular thrombus.
* Presence of a cardiac tumor.
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2008-09; Primary Completion 2009-06 (Estimated); Study Completion 2010-02 (Estimated)

PRIMARY OUTCOMES:
Safety, Adverse Events | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Grimm, Prof. MD, Principal Investigator — Vienna General Hospital, Clinical department for Cardiothoracic Surgery, Währinger Gürtel 18-20,1090 Vienna, Austria
Locations (1):
- Clinical Department for Cardiothoracic Surgery, General Hospital Vienna, Vienna, Austria